CLINICAL TRIAL: NCT04372459
Title: Online Psychosocial Cancer Screening, Monitoring and Stepped Treatment in Cancer Survivors: A Randomized Controlled Trial
Brief Title: Online Psychosocial Cancer Screening, Monitoring and Stepped Treatment in Cancer Survivors
Acronym: ICOnnectat-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Cristian Ochoa Arnedo, PhD, Clinical Psychologist, Institut Català d'Oncologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICOnnectat-BC; PI19/01880 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Psychological Distress; Emotional Disorder
Keywords: e-health; breast cancer; survivors; psychosocial care; distress; Randomised Controlled Trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The current clinical trial is a multicenter Randomised Controlled Trial with 2 parallel groups. The effectiveness of the online integrated and stepped psychosocial care group will be compared with the usual psychosocial care group
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online integrated and stepped psychosocial care (Experimental): A group of breast cancer survivors will be randomly allocated (1:1 allocation) to the online integrated and stepped psychosocial care group
  Interventions: Behavioral: Online integrated and stepped psychosocial care
- Usual psychosocial care (Experimental): A group of breast cancer survivors will be randomly allocated (1:1 allocation) to the usual psychosocial care group
  Interventions: Behavioral: Usual psychosocial care

INTERVENTIONS:
Behavioral: Online integrated and stepped psychosocial care — This program features four levels of care, increasing in intensity of psychosocial care as patients move from one level to the next one.
  Step 1: Screening and monitoring of several psychosocial variables through the central mobile application of the program (App ICOnnecta't).
  Step 2: Online guided and self-help psychoeducation Campus in which patients can consult videos and online resources, co-constructed between health professionals and patients, containing reliable and rigorous information related to the oncological process.
  Step 3: Online community of psychosocial support. Participants can choose from 12 cancer-related discussion forums and share with the community any health-related question that worries them fostering, thus, debate and stimulating peer-support.
  Step 4: Intensive online group psychotherapy (App ICOnnecta't Videoconsultation), based on the Group Positive Psychotherapy program for cancer survivors (Ochoa, Sumalla, Maté, Castejón, Rodríguez et al., 2010).
  Arms: Online integrated and stepped psychosocial care
Behavioral: Usual psychosocial care — This active control group will receive the standard psychosocial treatment for cancer survivors in the participating centers, led by a clinical psychologist and consisting of 8 individual, 45/60-minute sessions, each of which every 1-2 months, focused on providing emotional support and psychoeducation during the first year of primary cancer treatment.
  Arms: Usual psychosocial care

SUMMARY:
This multicenter randomized controlled study will appraise the effectiveness and cost-utility of an e-health ecosystem with integrated and stepped psychosocial services that will be compared with the usual psychosocial care. The study is developed in the acute survival phase among breast cancer survivors. The outcomes of both interventions will be compared in terms of the amount of waiting time to receive psychosocial care and changes in several psychosocial variables. Finally, a comparative economic analysis will be conducted in other relevant psychosocial and health parameters. The e-health platform is expected to outperform usual care in the aforementioned indicators, while reaching high acceptability and usability by survivors, and additionally reducing costs for health providers.

DETAILED DESCRIPTION:
Cancer diagnosis and treatment causes a huge psychosocial impact on breast cancer survivors. Psychosocial treatments in cancer survivors have already demonstrated their effectiveness in reducing emotional distress and improving quality of life although the access to them still presents important barriers, such as poor early detection, long waiting times for diagnosis or treatment, as well as other restrictions related to work, mobility or economic situation. In addition, the current digitization of screening, monitoring and psychosocial treatment poses a revolution in the improvement of the quality of care and the reduction of its economic burden. The objectives of this study are, first, to assess the clinical efficacy of an e-health platform that includes integrated and stepped psychosocial services, in comparison to usual psychosocial care, and second, to examine its cost-utility.

The study methodology is that of a multicentre randomised controlled trial with 2 parallel groups (experimental versus control group). Approximately 193 patients diagnosed with breast cancer in the acute survival phase will be recruited from 3 University hospitals in Catalonia (Spain) and will be randomised to one of two treatment conditions. All participants will be evaluated at the beginning of the study (T1: recruitment), 3 months from T1 (T2), 6 months from T1 (T3) and 12 months from T1 (T4). Primary outcome measures will include detection of clinical cases, amount of waiting time from detection to psychosocial intervention, and proportion of cases solved in the different steps of the intervention, as well as outcomes related to emotional distress, quality of life, post-traumatic stress and growth and therapeutic alliance. Secondary outcomes will include the acceptability of the platform by patients through satisfaction questionnaires and the usability of the platform. For the cost-utility analysis, the investigators will assess quality-adjusted life years (QALYs) and costs related to the number of days of sick leaves, healthcare utilization, adherence to pharmacological treatment, health professionals' costs, infrastructure and transport costs.

The study will provide an important advance in the treatment of breast cancer; in the long term, it is expected to improve the quality of patient care and the treatment efficacy and to reduce waiting lists as well as direct and indirect costs associated with the treatment of the disease in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years with BC, within 6 weeks after diagnosis.
* Having online access and a user-level knowledge of Internet.
* Understanding of Spanish language.

Exclusion Criteria:

* Major depressive episode.
* Significant autolytic ideation.
* Showing symptoms of psychosis or substance abuse.
* Intellectual disability.
* Having a mobile phone with an old release of Android operating system, which is not compatible with the platform.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Distress (HADS) | Time 1: Baseline; Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983; Spanish validation by Costa-Requena, Pérez Martín, Salamero Baró, & Gil Moncayo, 2009). It consists of 14 items, 7 for anxiety and 7 for depression, on a four-point Likert scale (range 0-3), with the total score ranging from 0 to 42. Higher scores indicate a greater level of distress.
Change in Post-traumatic Stress (PCL-5) | Time 1: Baseline; Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  Post-traumatic Stress Disorder Checklist-Civilian version (PCL-5) (Blevins, Weathers, Davis, Witte, & Domino, 2015). The official Spanish translation of the instrument was provided by the National Center for Post-Traumatic Stress Disorder (www.ptsd.va.gov/). The PCL-5 is a 20-item questionnaire, corresponding to the "Diagnostic and Statistical Manual for Mental Disorders Version 5" symptom criteria for PTSD. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items, with higher scores indicating worse outcomes.
Change in Post-traumatic Growth (PTGI) | Time 1: Baseline; Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  Post-traumatic Growth Inventory (PTGI) (Tedeschi & Calhoun, 1996; Spanish validation by Costa-Requena and Gil, 2007). It is a 21-item instrument based on a 6-point Likert scale (0=no change - 5=very high degree of change), which assesses positive changes experienced after a trauma. Total scores range from 0 to 105 with higher scores indicating better outcomes.
Change in Therapeutic alliance (WAI-P) | Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  Working Alliance Inventory-Patient Version (WAI-P; Horvath, 1981; Horvath & Greenberg, 1986, 1989; Spanish validation by Andrade-González & Fernández-Liria, 2015). It consists of 36 items with seven possible response options (1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always). The scoring range of the overall WAI-P is 36-252 points with higher scores indicating better outcomes.
Change in Quality of Life (EQ-5D-3L) | Time 1: Baseline; Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  EuroQoL-EQ-5D-3L (EuroQol Group, 1990; Spanish validation by Abadia et al., 1999). It consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Total scores range from 0-100 with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Healthcare utilization | Time 4: 12 months post-intervention
  Total number of visits to each healthcare professional (oncologist, nursing staff, psychologist, psychiatrist, social worker, emergency department) (Electronic Health Record).
Change in Medication use and adherence (ARMS) | Time 1: Baseline; Time 2: Change between Time 1 and 3 months post-intervention; Time 3: Change between Time 1 and 6 months post-intervention; Time 4: Change between Time 1 and 12 months post-intervention
  Adherence to Refills and Medications Scale (ARMS; Kripalani, Risser, Gatti, & Jacobson, 2009; Spanish validation by Gonzalez-Bueno et al., 2017). It consists of 12 questions: 8 aimed at assessing the patient's ability to properly administer the medication and 4 regarding its correct intake based on a four-point Likert scale (range from 1=never to 4=always; total score range 12-48), with lower scores indicating better adherence.
Work absenteeism | Time 4: 12 months post-intervention
  Number of days of patients' sick leaves (Electronic Health Record).
Professionals' salaries | Time 4: 12 months post-intervention
  Number of professionals involved in the online treatment or usual care as well as the number of professionals' working hours per week and costs (Electronic Health Record).
Infrastructure costs | Time 4: 12 months post-intervention
  Costs per user and per month for the development and maintenance of the online platform (experimental group) and costs of hospital's infrastructure per face-to-face visits per user and month.
Transport costs | Time 4: 12 months post-intervention
  Cost estimate per patient using a specific transport according to mobility data in Catalonia area.

OTHER OUTCOMES:
Emotional wellbeing (experimental group only) | Administration every 7 days until the end of treatment (or study completion), an average of 1 year
  Emotional thermometer (ET) - Visual Analogue Scale (VAS) (0-10) of the ICOnnecta't application.
Health education | Single administration per educational topic (7 thematic blocks, 16 topics, 40 questionnaires) until the end of treatment (or study completion), an average of 1 year
  Scores on health education questionnaires from Campus of ICOnnecta't. Higher scores indicate better health education acquisition.
Usability (experimental group only) (SUS) | 21 days after registration
  System Usability Scale (SUS) (Brooke, 1996). The SUS is a 10-item questionnaire with five response options that range from 4 = "Strongly agree" to 0 = "Strongly disagree". The SUS provides a "quick and dirty" reliable tool for measuring the usability of a range of systems.The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Higher scores indicate better outcomes.
Satisfaction (experimental group only) | 21 days after registration
  Visual Analogue Scale (VAS) (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Ochoa, PhD, Principal Investigator — Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain, 08908
Locations (1):
- Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The following IPD are to be shared with other researchers: Age (aggregated), civil status (aggregated), education (aggregated), occupational status (aggregated), date of enrolment (aggregated), date of opt out (aggregated and if applicable), date of oncological diagnosis (aggregated), cancer stage, oncological treatment (aggregated), psychotropic medication (aggregated), treatment arm in the study, and results from scales and subscales of psychometric instruments. Only ITT participants' data will be retained in the dataset.
Supporting Information: Study Protocol
Time Frame: January 2023-January 2033
Access Criteria: Access will be granted through formal requests from interested researchers. In order to keep control on data access we will register contact details of these scientists and their objectives for data use.

REFERENCES:
- [Derived] Ochoa-Arnedo C, Medina JC, Flix-Valle A, Anastasiadou D. E-health ecosystem with integrated and stepped psychosocial services for breast cancer survivors: study protocol of a multicentre randomised controlled trial. BMJ Open. 2021 Mar 8;11(3):e041548. doi: 10.1136/bmjopen-2020-041548. PMID 34006024